CLINICAL TRIAL: NCT00951457
Title: Bendamustine Combined With Alemtuzumab in Pretreated Chronic Lymphocytic Leukemia (CLL) - A Phase I/II Trial With Concomitant Evaluation of Safety and Efficacy
Brief Title: Bendamustine Combined With Alemtuzumab in Pretreated Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Mundipharma Pte Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT CLL-6 BendAlem
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2017-12

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: CLL; pretreated; immune therapy; dose escalation; maintenance therapy; Bendamustine; Alemtuzumab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Overall study (Experimental): Dose escalation phase:
  Days -3, -2, -1: 3 - 10 - 30 mg Alemtuzumab s.c.
  Treatment phase:
  Bendamustine 70 mg/m2 i.v. on d1 + d2 repeat every 28 days for 4 cycles
  Alemtuzumab 30 mg s.c. 3x per week (days 1, 3, 5) continuously in parallel with chemotherapy cycles for a maximum of 16 weeks
  Interventions: Drug: Bendamustine; Drug: Alemtuzumab

INTERVENTIONS:
Drug: Bendamustine
  Other Names: Ribomustin
Drug: Alemtuzumab

SUMMARY:
The primary objective of this study is to determine the percentage of patients achieving a response, defined as the percentage of patients achieving complete response, partial response and stable disease/ no change upon treatment with the combination therapy according to NCI response criteria (also established according to IWCLL guidelines) upon treatment with a combination of bendamustine and alemtuzumab.

DETAILED DESCRIPTION:
This is a non-randomized, multicenter, open-label, single-arm Phase I/II study to evaluate the safety and efficacy of bendamustine combined with alemtuzumab in patients with pretreated CD20-positive CLL (according to the revised NCI/ IWCLL criteria).

Eligible patients will receive bendamustine as 4 courses of 70 mg/m2 on days 1 and 2 every 28 days and 30 mg alemtuzumab s.c. continuously on days 1, 3 and 5 of every week, for a maximum of 16 weeks. Safety assessments will be conducted weekly; efficacy assessments including imaging will be performed at months 2, 4, 6, 10 and 16. Bone marrow biopsies will be performed upon CR (according to the 2008 IWCLL response criteria) or fixed at 6 and 16 months.

Following recruitment of the first 3 and 7 patients safety evaluations will be performed by a data safety monitoring board. An interim analysis for response and safety as well as maximum tolerated dose levels will occur after the first 7 patients have completed treatment (Gehan timepoint). If the treatment is deemed clinically safe a further 13 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with CD23+, CD5+, CD19+ light chain monoclonal B-CLL with treatment indication according to IWCLL criteria (Appendix 4)
* 1st or greater relapse after fludarabine or any other primary treatment regimen OR Refractory to any previous treatment and simultaneous indication for treatment according to IWCLL criteria (Appendix 4)
* Age 18 years and older
* ECOG status 0 - 2
* Life expectancy > 6 months
* Written informed consent given by the patient
* Patient using a reliable means of contraception (e.g. physical barrier, contraceptive pill or patch, spermicide and barrier, or IUD) for the duration of the study. Male patients have to use an adequate contraception method for the duration of study treatment and for 6 months following completion of study treatment. Women of childbearing potential have to use an effective method of contraception for the duration of study participation.

Exclusion Criteria:

* HIV positive or positive for Hepatitis B or C
* Active uncontrolled infection
* Pregnant or lactating women
* Hypersensitivity with anaphylactic reaction to humanised monoclonal antibodies or to the excipients of any of the applied drugs (e.g. Bendamustine hydrochloride or mannitol)
* Previous treatment with bendamustine
* Treatment with an experimental drug within the previous 2 months
* Patients with a history of other malignancies within 2 years prior to study entry, except for adequately treated carcinoma in situ of the cervix; basal or squamous cell skin cancer; low grade, early stage localized prostate cancer treated surgically with curative intent; good prognosis DCIS of the breast treated with lumpectomy alone with curative intent.
* Transformation to aggressive B-cell malignancy (e.g. large B-cell lymphoma, Richter's syndrome, or prolymphocytic leukemia (PLL)
* Decreased kidney function with creatinine clearance < 30 ml/min
* Patients with severe co-morbidities or major organ dysfunctions (e.g. known severe liver damage, jaundice)
* Patients with a history of severe cardiac disease; e.g. NYHA Functional Class III or IV heart failure, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, or unstable angina
* Any co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent, or patients unable to comply with requirements of study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2012-08-06 (Actual); Study Completion 2012-08-06 (Actual)

PRIMARY OUTCOMES:
To determine the percentage of patients achieving a response, defined as the percentage of patients achieving complete response, partial response and stable disease/ no change upon treatment with the combination therapy | 2 -16 months

SECONDARY OUTCOMES:
To evaluate the efficacy of a bendamustine/ alemtuzumab combination therapy in terms of complete response rates | 2 - 16 months
To evaluate the achievable cumulative doses of bendamustine and alemtuzumab in terms of maximum tolerated doses while on treatment | 2 -16 months
To determine response rates in all phases by 4-colour flow cytometric MRD analysis | 2 -16 months
To identify and characterize potential risk factors via FISH cytogenetics, CD38/ Zap-70 expression and mutational status | 2 - 6 months
To define clonal evolution by use of longitudinal FISH cytogenetics | 2 - 6 months
To define T cell subsets including prognostic EM T cells and Treg cells | 2 - 16 months
To document change upon quality of life by use of a standardized QoL questionnaire | 2 -16 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, Prof.Dr., Study Chair — Arbeitsgemeinschaft medikamentoese Tumortherapie
Locations (7):
- Austria (7):
  - Medizinische Universitaet Innsbruck, Abtlg. f. Haematologie und Onkologie, Innsbruck, Tyrol
  - Landeskrankenhaus Feldkirch, Feldkirch
  - A.ö. Landeskrankenhaus Leoben, Leoben
  - Krankenhaus der Elisabethinen Linz, Linz
  - Krankenhaus der Stadt Linz, Linz
  - Universitaetsklinik f. Innere Medizin III, Salzburg
  - Klinikum Wels-Grieskirchen GmbH, Wels